CLINICAL TRIAL: NCT01746004
Title: Disposition of [14C]-LY2157299 Monohydrate Following Oral Administration in Healthy Subjects
Brief Title: A Study of LY2157299 Monohydrate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14671; H9H-MC-JBAM (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [^14C]-LY2157299 (Experimental): Single 150 mg oral dose of LY2157299 monohydrate containing 100 micro curies of [^14C] labeled drug
  Interventions: Drug: [^14C]-LY2157299

INTERVENTIONS:
Drug: [^14C]-LY2157299 — [^14C]-LY2157299 monohydrate administered as oral solution

SUMMARY:
This study involves a single dose of 150 milligram (mg) of radiolabeled LY2157299 monohydrate in healthy participants. The study will determine how the body eliminates the radioactivity and LY2157299 monohydrate. Participants must be healthy surgically sterile or postmenopausal females, or sterile males. This study is approximately 8 to 15 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy surgically sterile females, postmenopausal females, or sterile males
* Body mass index (BMI) of 18.5 to 32.0 kilograms per square meter (kg/m^2)
* Have venous access sufficient to allow for blood sampling

Exclusion Criteria:

* Have known allergies to LY2157299, related compounds or any components of the formulation
* Have an abnormal blood pressure as determined by the investigator
* Have participated in a [^14C]-study within the last 6 months prior to admission for this study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Urinary and Fecal Excretion of LY2157299 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Pre-dose through Day 15

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of LY2157299 and Radioactivity Maximum Observed Concentration (Cmax) | Pre-dose through Day 14
Plasma Pharmacokinetics (PK) of LY2157299 and Radioactivity Time of Maximum Observed Concentration (Tmax) | Pre-dose through Day 14
Plasma Pharmacokinetics (PK) of LY2157299 and Radioactivity Area Under the Concentration-Time Curve from Time Zero to the Last Timepoint with a Measurable Concentration (AUC 0 to tlast) | Pre-dose through Day 14
Relative Abundance of LY2157299 and the Metabolites of LY2157299 in Urine and Feces | Pre-dose through Day 14
Relative Abundance of LY2157299 and the Metabolites of LY2157299 in Plasma | Pre-dose through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin, United States